CLINICAL TRIAL: NCT01712074
Title: A Randomized, 18-week, Placebo-controlled, Double-blind, Parallel Group Study Of The Safety And Efficacy Of Pf-05212377 (Sam-760) In Subjects With Mild-to-moderate Alzheimer's Disease With Existing Neuropsychiatric Symptoms On A Stable Daily Dose Of Donepezil
Brief Title: Study Evaluating TheSafety And Efficacy Of PF-05212377 Or Placebo In Subjects With Alzheimer's Disease With Existing Neuropsychiatric Symptoms On Donepezil
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated October 23, 2015 as pre-specified, interim analysis futility criteria were met. The termination was not due to safety concerns.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B2081011; 2014-000830-42 (EudraCT Number)
Record Dates: First submitted 2012-10-19; First posted 2012-10-23 (Estimated); Results first posted 2017-03-20 (Actual); Last update posted 2017-03-20 (Actual); Status verified 2017-01

CONDITIONS: Alzheimer's Disease
Keywords: Randomized; Double Blind; Safety and Efficacy
MeSH Terms: conditions — Alzheimer Disease | interventions — SAM-760

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 30 mg QD of PF-05212377 (Experimental)
  Interventions: Drug: PF-05212377 (SAM-760)
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: PF-05212377 (SAM-760) — 30 mg QD of PF-05212377 (SAM-760)
  Arms: 30 mg QD of PF-05212377
Other: Placebo — Placebo QD
  Arms: Placebo

SUMMARY:
This study will evaluate safety and efficacy of PF-05212377 in subjects with mild-to-moderate Alzheimer's Disease with existing neuropsychiatric symptoms on a stable dose of Donepezil. The 4-week run-in will minimize placebo effect. The 12-week treatment period is considered the minimum length necessary to reliably evaluate the effect PF-05212377 on cognition and and neuropsychiatric symptoms in this population. The 2-week washout will allow to monitor re-emergence of neuropsychiatric and cognitive symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of probable AD with supportive brain imaging documentation
* Have existing neuropsychiatric symptoms as defined by a score equal or greater than 10 on the NPI at screening, arising from item scores equal or greater than 2 (frequency X severity) on at least 2 domains.
* Has been on donepezil (stable dose of 5 mg or 10 mg) for at least four months, with no intent to change such for the duration of the study.

Exclusion Criteria:

* Demonstrate extreme agitation, physical aggression or violence to themselves, their caregiver, or others, and/or an inability to complete the ADAS-cog assessment at Screening.
* Have major structural brain disease other than Alzheimer's Disease
* Other severe acute or chronical medical or psychiatric condition or laboratory abnormality

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2012-11; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (60):
- United States (40):
  - ATP Clinical Research, Inc, Costa Mesa, California
  - Sun Valley Research Center, Imperial, California
  - Desert Valley Research, Rancho Mirage, California
  - RAA - Apex Aquisition, LLC, Santa Ana, California
  - Geriatric and Adult Psychiatry LLC, Hamden, Connecticut
  - Yale University, New Haven, Connecticut
  - Yale-New Haven Hospital, Temple Radiology, New Haven, Connecticut
  - Yale University School of Medicine, MRI Research Center (MRI), New Haven, Connecticut
  - Diagnostic Centers of America, Boynton Beach, Florida
  - Meridien Research, Brooksville, Florida
  - Quantum Laboratories, Deerfield Beach, Florida
  - Brain Matters Research Inc, Delray Beach, Florida
  - MD Clinical, Hallandale, Florida
  - Compass Research LLC-North Clinic, Leesburg, Florida
  - Medical Research Group of Central Florida, Orange City, Florida
  - Premiere Research Institute, West Palm Beach, Florida
  - Institute for Advanced Medical Research, Alpharetta, Georgia
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - Columbus Research & Wellness Institute, Inc., Columbus, Georgia
  - Lake Charles Clinical Trials, Lake Charles, Louisiana
  - Michigan State University, East Lansing, Michigan
  - Metro Imaging (Imaging only), Creve Coeur, Missouri
  - Millennium Psychiatric Associates, LLC, Creve Coeur, Missouri
  - Eastside Comprehensive Medical Center, LLC, New York, New York
  - University of Rochester Medical Center AD-CARE Program | University of Rochester Medical Center, Rochester, New York
  - University of Rochester Medical Center (MRI Imaging Only), Rochester, New York
  - Behavioral Medical Research of Staten Island, Staten Island, New York
  - The Ohio State University (administrative offices only), Columbus, Ohio
  - The Ohio State University - 2050, Columbus, Ohio
  - Keystone Clinical Studies, LLC, Norristown, Pennsylvania
  - Roper Hospital (Imaging Only), Charleston, South Carolina
  - Roper St. Francis Healthcare, Charleston, South Carolina
  - Roper St. Francis Pharmacy (IP Shipment/Storage), Charleston, South Carolina
  - Neurology Clinic, P.C., Cordova, Tennessee
  - Senior Adults Speciality Research Inc., Austin, Texas
  - Grayline Clinical Drug Trials, Wichita Falls, Texas
  - Clinical Neuroscience Research Assoc. d/b/a The Memory Clinic, Bennington, Vermont
  - Dean Foundation for Health, Research and Education, Middleton, Wisconsin
  - Cary J. Kohlenberg, MD, dba, IPC Research, Waukesha, Wisconsin
  - Merrill Hills Manor, Waukesha, Wisconsin
- Canada (4):
  - True North Clinical Research Halifax, Inc., Halifax, Nova Scotia
  - Chatham-kent Clinical Trials Research Centre, Chatham, Ontario
  - Chatham-Kent Clinical Trials Research Centre, Chatham, Ontario
  - Recherches Neuro-Hippocampe Inc., Gatineau, Quebec
- Chile (3):
  - Psicomed Estudios Medicos CIA. LTDA, Antofagasta, Antofagasta
  - Biomedica Research Group, Santiago, Santiago Metropolitan
  - Especialidades Medicas L Y S, Santiago, Santiago Metropolitan
- Espace Sante 2, La Seyne-sur-Mer, France
- Germany (5):
  - Dr. med. Volker Schumann, Arzt fuer Nervenheilkunde, Berlin
  - Praxis Dr. Franz- Arztehaus am KEH mit Epilepsie-Zentrum, Berlin
  - Praxis Dr. sc. med. Alexander Schulze, Berlin
  - Arzneimittelforschung Leipzig Gmbh, Leipzig
  - Praxis fuer Neurologie / Psychiatrie Prof. Dr. Steinwachs, Nuremberg
- Spain (2):
  - Hospital General Universitario De Elche, Elche, Alicante
  - Hospital de Cantoblanco, Madrid, Madrid
- United Kingdom (5):
  - The Research Institute for the Care of Older People Centre, Bath
  - Fulbourn Hospital, Cambridge
  - Surrey and Borders Partnership NHS Foundation Trust, Chertsey
  - Berrywood Hospital, Northampton
  - Covance Laboratories, Switzerland

REFERENCES:
- [Derived] Fullerton T, Binneman B, David W, Delnomdedieu M, Kupiec J, Lockwood P, Mancuso J, Miceli J, Bell J. A Phase 2 clinical trial of PF-05212377 (SAM-760) in subjects with mild to moderate Alzheimer's disease with existing neuropsychiatric symptoms on a stable daily dose of donepezil. Alzheimers Res Ther. 2018 Apr 5;10(1):38. doi: 10.1186/s13195-018-0368-9. PMID 29622037
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B2081011&StudyName=Study%20Evaluating%20TheSafety%20And%20Efficacy%20Of%20PF-05212377%20Or%20Placebo%20In%20Subjects%20With%20Alzheimer%27s%20Disease%20With%20Existing%20Neuropsychiatric%20Symp

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Before entering in the 12-week treatment period, participants were required to enter a 4-week placebo run-in period. 195 participants started the placebo run-in period, of which 186 were eligible for the treatment period. Among the 186 enrolled participants, 185 were treated with the double-blind study treatment, 1 was enrolled but not treated.
Pre-assignment Details: This study was a multicenter Phase 2a, randomized, placebo controlled, safety and efficacy study of 18 weeks in duration in participants with mild-to-moderate Alzheimer's disease (AD) who were stable on treatment with 5 or 10 mg of donepezil and who had existing neuropsychiatric symptoms.
Groups:
- Placebo Run-In: Participants that received placebo during the 4-week single blind placebo run-in period
- PF-05212377 30 mg: Double Blind Period: All participants that received PF-05212377 30 mg during the 12-week double blind period
- Placebo: Double Blind Period: All participants that received placebo during the 12-week double blind period
Period: Placebo Run-in Period
Arm/Group | Placebo Run-In | PF-05212377 30 mg: Double Blind Period | Placebo: Double Blind Period
Started | 195 | 0 | 0
Completed | 185 | 0 | 0
Not Completed | 10 | 0 | 0
Not completed — Adverse Event | 2 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — No longer meets eligibility criteria | 5 | 0 | 0
Not completed — Other | 1 | 0 | 0
Not completed — No longer willing to participate | 1 | 0 | 0
Period: Double Blind Period
Arm/Group | Placebo Run-In | PF-05212377 30 mg: Double Blind Period | Placebo: Double Blind Period
Started | 0 | 91 | 94
Completed | 0 | 77 | 86
Not Completed | 0 | 14 | 8
Not completed — Adverse Event | 0 | 2 | 1
Not completed — No longer willing to participate | 0 | 2 | 4
Not completed — Death | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 2 | 1
Not completed — Other | 0 | 4 | 1
Not completed — Protocol Violation | 0 | 0 | 1
Not completed — No longer met eligibility criteria | 0 | 3 | 0

BASELINE CHARACTERISTICS:
Population: One (1) of participant randomized but not treated appeared under placebo run-in including his/her discontinued and safety information
Groups:
- Not Randomized: Participants who have been discontinued during the Placebo Run-In period
- PF-05212377 30 mg: Double Blind Period: All participants entered the double blind period and received PF-05212377 30 mg
- Placebo: Double Blind Period: All participants entered the double blind period and received placebo
- Total: Total of all reporting groups
Arm/Group | Not Randomized | PF-05212377 30 mg: Double Blind Period | Placebo: Double Blind Period | Total
Number analyzed (Participants) | 9 | 92 | 94 | 195
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.2 (8.8) | 76.0 (8.0) | 75.9 (7.5) | 76 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  FEMALE | 7 | 46 | 55 | 108
  MALE | 2 | 46 | 39 | 87

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in ADAS-cog13 Total Score at Week 16
Description: ADAS-cog13 (13-item ADAS cog) is a psychometric instrument that evaluates word recall, ability to follow commands, constructional praxis, naming, ideational praxis, orientation, word recognition, memory, comprehension of spoken language, word-finding, and language ability, with a measure of delayed word recall and concentration/ distractibility. The total score of the 13-item scale ranges from 0 to 85, with an increase in score indicating cognitive worsening.
Time Frame: Baseline and Week 16
Population: The Full Analysis Set (FAS) is defined as all participants who were randomized. The FAS was the primary analysis set for efficacy data.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Groups:
- PF-05212377 30 mg: participants who received PF-05212377 30 mg contributing to the analysis during double blind period
- Placebo: All participants who received placebo contributing to the analysis during the double blind period
Arm/Group | PF-05212377 30 mg | Placebo
Number analyzed (Participants) | 78 | 86
scores on a scale | 0.111 (0.6290) | -0.584 (0.5995)
Statistical Analysis 1: Comparison: PF-05212377 30 mg vs Placebo; Test type: Superiority or Other; p = 0.4256, Mixed Models Analysis; Mean Difference (Net) = 0.695, 80% CI 2-sided [-0.424 to 1.814], Standard Error of Mean 0.8697

2. Secondary Outcome: Change From Baseline in the Neuropsychiatric Inventory (NPI) Total Score at Week 16 (Visit 5)
Description: The NPI evaluates both frequency and severity of 12 neuropsychiatric disturbances including delusions, hallucinations, agitation/aggression, depression/dysphoria, anxiety, elation/euphoria, apathy/indifference, disinhibition, irritability/lability, motor disturbance, nighttime behaviors, as well as appetite/eating. The NPI total score (for 12 behavioral domains) is calculated as the product of frequency and severity for each domain, and ranges from 0 to 144. An increase in score indicates a worsening of symptoms.
Time Frame: Baseline and Week 16
Population: The FAS is defined as all participants who are randomized. The FAS was the primary analysis set for efficacy data.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | PF-05212377 30 mg | Placebo
Number analyzed (Participants) | 78 | 87
scores on a scale | -3.990 (1.2441) | -6.184 (1.1801)
Statistical Analysis 1: Comparison: PF-05212377 30 mg vs Placebo; Test type: Superiority or Other; p = 0.2027, Mixed Models Analysis; Mean Difference (Net) = 2.194, 80% CI 2-sided [-0.013 to 4.401], Standard Error of Mean 1.7149

3. Other Pre Specified Outcome: Percentage of Participants With Treatment Emergent Adverse Events (TEAEs) Leading to Discontinuation
Description: Proportion of participants with TEAEs leading to discontinuation over the 12-week double blind treatment period and washout. Adverse events (AEs) occurring following start of treatment or increasing in severity were counted as treatment emergent
Time Frame: Week 4 to Week 18
Population: All participants who received any treatment during double blind period
Measure: Number; unit: Percentage of Participants
Groups:
- Placebo: All participants receiving placebo during double blind period
Arm/Group | PF-05212377 30 mg | Placebo
Number analyzed (Participants) | 91 | 94
Percentage of Participants | 3.3 | 0

4. Other Pre Specified Outcome: Proportion of Participants With Laboratory Abnormalities of Potential Clinical Concern During Double Blind Period
Description: Proportion (%) of participants with laboratory abnormalities (without regard to baseline abnormalities) of potential clinical concern over the 12-week double blind treatment period.
  The following laboratory parameters were analyzed: hematology (hemoglobin, hematocrit, red blood cell count, platelet count, white blood cell count, total neutrophils, eosinophils, monocytes, basophils, lymphocytes); blood chemistry (blood urea nitrogen, creatinine, glucose, calcium, sodium, potassium, chloride, total bicarbonate, aspartate aminotransferase, alanine aminotransferase, bilirubin, alkaline phosphatase, uric acid, albumin, and total protein; urinalysis (pH, glucose, protein/albumin, hemoglobin/blood, ketones/acetone, nitrites, leukocyte esterase, microscopy [if urine dipstick was positive for blood, protein, nitrites or leukocyte esterase]); others (only at screening or needed: urine drug screen, thyroid panel, Vitamin B12, methylmalonic acid, folate and Hemoglobin A1).
Time Frame: Week 4 to Week 16
Population: All participants who received any treatment during Week 4 (Visit 2) to Week 16 (Visit 5)
Measure: Number; unit: Percentage of Participants
Groups:
- Placebo: All participants receiving placebo with non-missing clinical laboratory data during double blind period
Arm/Group | PF-05212377 30 mg | Placebo
Number analyzed (Participants) | 91 | 94
Percentage of Participants | 36.0 | 52.0

5. Other Pre Specified Outcome: Selected ECG Change From Baseline - PR Interval at Week 6 (Visit 3)
Description: The PR interval is the time from the onset of the P wave to the start of the QRS complex (the combination of the Q wave, R wave and S wave, representing ventricular depolarization).
Time Frame: Baseline and Week 6
Population: All participants who received any treatment during Week 4 (Visit 2) to Week 16 (Visit 5)
Measure: Mean (Full Range); unit: milliseconds (msec)
Groups:
- Placebo: All participants who received placebo with non-missing ECG data during the double blind period
Arm/Group | PF-05212377 30 mg | Placebo
Number analyzed (Participants) | 85 | 89
milliseconds (msec) | -2.8 [-52 to 24] | -3.6 [-82 to 35]

6. Other Pre Specified Outcome: Selected ECG Change From Baseline - PR Interval at Week 10 (Visit 4)
Description: as for outcome 5
Time Frame: Baseline and Week 10
Population: All participants who received any treatment during Week 4 (Visit 2) to Week 16 (Visit 5)
Measure: Mean (Full Range); unit: msec
Groups:
- Placebo: All participants receiving placebo with non-missing ECG data during double blind period
Arm/Group | PF-05212377 30 mg | Placebo
Number analyzed (Participants) | 79 | 87
msec | -0.1 [-42 to 23] | -1.3 [-61 to 61]

7. Other Pre Specified Outcome: Selected ECG Change From Baseline - PR Interval at Week 16/Early Termination (Visit 5)
Description: as for outcome 5
Time Frame: Baseline and Week 16/Early Termination
Population: All participants who received any treatment during Week 4 (Visit 2) to Week 16 (Visit 5)
Measure: Mean (Full Range); unit: msec
Arm/Group | PF-05212377 30 mg | Placebo
Number analyzed (Participants) | 82 | 85
msec | -2.5 [-69 to 24] | -1.6 [-49 to 33]

8. Other Pre Specified Outcome: Percentage of Participant With PR Interval Abnormalities of Potential Clinical Concern
Description: Proportion (%) of participants with PR Interval abnormalities meeting categorical criteria over the 12 week double blind treatment period. The PR interval is the time from the onset of the P wave to the start of the QRS complex (the combination of the Q wave, R wave and S wave, representing ventricular depolarization). Participants with post-baseline PR absolute value>=300 msec , a PR increase of >=25% (for participants with a baseline value>=200 msec), or with an increase >=50% (for participants with a baseline value<200 msec) were counted.
Time Frame: Week 4 to Week 16
Population: All participants who received any treatment during Week 4 (Visit 2) to Week 16 (Visit 5)
Measure: Number; unit: Percentage of Participants
Arm/Group | PF-05212377 30 mg | Placebo
Number analyzed (Participants) | 86 | 90
Percentage of Participants
  Post-Baseline Maximum Absolute Value >=300 msec | 0 | 4.4
  Post-Baseline Maximum Increase >=25/50% | 0 | 0

9. Other Pre Specified Outcome: Selected ECG Change From Baseline - QRS Complex at Week 6 (Visit 3)
Description: The QRS complex is the combination of the Q wave, R wave and S wave, representing ventricular depolarization.
Time Frame: Baseline and Week 6
Population: All participants who received any treatment during Week 4 (Visit 2) to Week 16 (Visit 5)
Measure: Mean (Full Range); unit: msec
Arm/Group | PF-05212377 30 mg | Placebo
Number analyzed (Participants) | 88 | 92
msec | -0.3 [-22 to 43] | -0.8 [-14 to 10]

10. Other Pre Specified Outcome: Selected ECG Change From Baseline - QRS Complex at Week 10 (Visit 4)
Description: The QRS complex is the combination of the Q wave, R wave and S wave, representing ventricular depolarization.
Time Frame: Baseline and Week 10
Population: All participants who received any treatment during Week 4 (Visit 2) to Week 16 (Visit 5)
Measure: Mean (Full Range); unit: msec
Arm/Group | PF-05212377 30 mg | Placebo
Number analyzed (Participants) | 81 | 90
msec | -0.1 [-13 to 45] | 0.1 [-15 to 22]

11. Other Pre Specified Outcome: Selected ECG Change From Baseline - QRS Complex at Week 16/Early Termination (Visit 5)
Description: The QRS complex is the combination of the Q wave, R wave and S wave, representing ventricular depolarization.
Time Frame: Baseline and Week 16/Early Termination
Population: All participants who received any treatment during Week 4 (Visit 2) to Week 16 (Visit 5)
Measure: Mean (Full Range); unit: msec
Arm/Group | PF-05212377 30 mg | Placebo
Number analyzed (Participants) | 85 | 89
msec | 0.1 [-14 to 18] | -0.3 [-21 to 14]

12. Other Pre Specified Outcome: Proportion of Participants With QRS Complex Abnormalities of Potential Clinical Concern
Description: Proportion (%) of participants with QRS Complex abnormalities meeting categorical criteria over the 12 week double blind treatment period. The QRS complex is the combination of the Q wave, R wave and S wave, representing ventricular depolarization). Participants with post-baseline QRS complex absolute value>=100 msec , a QRS complex increase of >=25% (for participants with a baseline value>=100 msec), or with an increase >=50% (for participants with a baseline value<100 msec) were counted.
Time Frame: Week 4 to Week 16
Population: All participants who received any treatment during Week 4 (Visit 2) to Week 16 (Visit 5)
Measure: Number; unit: Percentage of participants
Arm/Group | PF-05212377 30 mg | Placebo
Number analyzed (Participants) | 91 | 93
Percentage of participants
  Post-Baseline Maximum Absolute Value >=200 msec | 0 | 0
  Post-Baseline Maximum Increase >=25/50% | 0 | 0

13. Other Pre Specified Outcome: Selected ECG Change From Baseline - QTcF Interval at Week 6 (Visit 3)
Description: The QTcF interval is a measure of the time between the start of the Q wave and the end of the T wave in the heart's electrical cycle, which is corrected for heart rate using Fridericia's formula.
Time Frame: Baseline and Week 6
Population: All participants who received any treatment during Week 4 (Visit 2) to Week 16 (Visit 5)
Measure: Mean (Full Range); unit: msec
Arm/Group | PF-05212377 30 mg | Placebo
Number analyzed (Participants) | 88 | 92
msec | -3.0 [-31 to 37] | -4.9 [-35 to 35]

14. Other Pre Specified Outcome: Selected ECG Change From Baseline - QTcF Interval at Week 10 (Visit 4)
Description: as for outcome 13
Time Frame: Baseline and Week 10
Population: All participants who received any treatment during Week 4 (Visit 2) to Week 16 (Visit 5)
Measure: Mean (Full Range); unit: msec
Arm/Group | PF-05212377 30 mg | Placebo
Number analyzed (Participants) | 81 | 90
msec | -0.2 [-38 to 47] | -5.5 [-40 to 48]

15. Other Pre Specified Outcome: Selected ECG Change From Baseline - QTcF Interval at Week 16/Early Termination (Visit 5)
Description: as for outcome 13
Time Frame: Baseline and Week 16/Early Termination
Population: All participants who received any treatment during Week 4 (Visit 2) to Week 16 (Visit 5)
Measure: Mean (Full Range); unit: msec
Arm/Group | PF-05212377 30 mg | Placebo
Number analyzed (Participants) | 85 | 89
msec | 0.8 [-31 to 34] | -2.2 [-62 to 30]

16. Other Pre Specified Outcome: Proportion of Participants With QTcF Interval Abnormalities of Potential Clinical Concern
Description: Proportion (%) of participants with QTcF Interval abnormalities meeting categorical criteria over the 12-week double blind treatment period. The QTcF interval is a measure of the time between the start of the Q wave and the end of the T wave in the heart's electrical cycle, which is corrected for heart rate using Fridericia's formula.
  Participants with a post-baseline QTcF absolute value of 450 - <480, 480 - <500, or >=500 mec, or with a post-baseline QTcF increase of 30 - <60 or >=60 msec were counted.
Time Frame: Week 4 to Week 16
Population: All participants who received any treatment during Week 4 (Visit 2) to Week 16 (Visit 5)
Measure: Number; unit: Percentage of Participants
Arm/Group | PF-05212377 30 mg | Placebo
Number analyzed (Participants) | 91 | 93
Percentage of Participants
  Post-Baseline Absolute Value of 450-<480 msec | 15.4 | 14.0
  Post-Baseline Absolute Value of 480-<500 msec | 4.4 | 1.1
  Change from Baseline of 30 -<60 msec | 6.6 | 3.2
  Change from Baseline >=60 msec | 0 | 0

17. Other Pre Specified Outcome: Blood Pressure (BP) Changes From Baseline - Week 6 (Visit 3)
Description: The BP changes from baseline at Week 6 (Visit 3) including supine systolic BP, standing systolic BP, standing systolic BP, supine diastolic BP, standing diastolic BP.
Time Frame: Baseline and Week 6
Population: All participants who received any treatment during Week 4 (Visit 2) to Week 16 (Visit 5)
Measure: Mean (Full Range); unit: millimeters of mercury (mm Hg)
Groups:
- Placebo: All participants receiving placebo with non-missing vital signs data during double blind period
Arm/Group | PF-05212377 30 mg | Placebo
Number analyzed (Participants) | 89 | 93
millimeters of mercury (mm Hg)
  Supine Systolic BP | -3.6 [-38 to 19] | -3.9 [-52 to 30]
  Standing Systolic BP | -4.1 [-49 to 20] | -3.0 [-38 to 22]
  Supine Diastolic BP | -2.2 [-37 to 26] | -1.8 [-33 to 20]
  Standing Diastolic BP | -1.1 [-23 to 17] | -1.0 [-23 to 21]

18. Other Pre Specified Outcome: Pulse Rate Changes From Baseline - Week 6 (Visit 3)
Description: The pulse rate changes from baseline at Week 6 (Visit 3) including supine pulse rate, and standing pulse rate.
Time Frame: Baseline and Week 6
Population: All participants who received any treatment during Week 4 (Visit 2) to Week 16 (Visit 5)
Measure: Mean (Full Range); unit: beats per minute (bpm)
Arm/Group | PF-05212377 30 mg | Placebo
Number analyzed (Participants) | 89 | 93
beats per minute (bpm)
  Supine Pulse Rate | -1.4 [-30 to 30] | 1.4 [-21 to 20]
  Standing Pulse Rate | -0.3 [-20 to 30] | 1.3 [-12 to 27]

19. Other Pre Specified Outcome: BP Changes From Baseline - Week 10 (Visit 4)
Description: The BP changes from baseline at Week 10 (Visit 4) including supine systolic BP, standing systolic BP, standing systolic BP, supine diastolic BP, standing diastolic BP.
Time Frame: Baseline and Week 10
Population: All participants who received any treatment during Week 4 (Visit 2) to Week 16 (Visit 5)
Measure: Mean (Full Range); unit: mmHg
Arm/Group | PF-05212377 30 mg | Placebo
Number analyzed (Participants) | 81 | 91
mmHg
  Supine Systolic BP | -3.4 [-36 to 20] | -0.3 [-68 to 34]
  Standing Systolic BP | -3.8 [-33 to 32] | 0.8 [-49 to 49]
  Supine Diastolic BP | -2.4 [-32 to 20] | -0.7 [-39 to 25]
  Standing Diastolic BP | -1.2 [-20 to 20] | 0.3 [-26 to 39]

20. Other Pre Specified Outcome: Pulse Rate Changes From Baseline - Week 10 (Visit 4)
Description: The pulse rate changes from baseline at Week 10 (Visit 4) including supine pulse rate, and standing pulse rate.
Time Frame: Baseline and Week 10
Population: All participants who received any treatment during Week 4 (Visit 2) to Week 16 (Visit 5)
Measure: Mean (Full Range); unit: bpm
Arm/Group | PF-05212377 30 mg | Placebo
Number analyzed (Participants) | 81 | 91
bpm
  Supine Pulse Rate | -0.4 [-26 to 22] | 0.5 [-24 to 17]
  Standing Pulse Rate | -0.7 [-20 to 24] | 1.8 [-19 to 21]

21. Other Pre Specified Outcome: BP Changes From Baseline - Week 16/Early Termination (Visit 5)
Description: The BP changes from baseline at Week 16/Early Termination (Visit 5) including supine systolic BP, standing systolic BP, standing systolic BP, supine diastolic BP, standing diastolic BP.
Time Frame: Baseline and Week 16/Early Termination
Population: All participants who received any treatment during Week 4 (Visit 2) to Week 16 (Visit 5)
Measure: Mean (Full Range); unit: mmHg
Arm/Group | PF-05212377 30 mg | Placebo
Number analyzed (Participants) | 85 | 90
mmHg
  Supine Systolic BP | -1.4 [-30 to 27] | -1.1 [-30 to 72]
  Standing Systolic BP | -1.0 [-30 to 32] | -1.1 [-26 to 66]
  Supine Diastolic BP | -2.1 [-39 to 22] | -0.3 [-18 to 35]
  Standing Diastolic BP | -0.8 [-23 to 23] | 0.0 [-20 to 36]

22. Other Pre Specified Outcome: Pulse Rate Changes From Baseline - Week 16/Early Termination (Visit 5)
Description: The pulse rate changes from baseline at Week 16/Early Termination (Visit 5) including supine pulse rate, and standing pulse rate.
Time Frame: Baseline and Week 16/Early Termination
Population: All participants who received any treatment during Week 4 (Visit 2) to Week 16 (Visit 5)
Measure: Mean (Full Range); unit: bpm
Arm/Group | PF-05212377 30 mg | Placebo
Number analyzed (Participants) | 85 | 90
bpm
  Supine Pulse Rate | -0.8 [-29 to 31] | 0.6 [-22 to 20]
  Standing Pulse Rate | -1.9 [-24 to 29] | 0.8 [-17 to 17]

23. Other Pre Specified Outcome: Proportion of Participants With Post-Baseline Vital Signs Abnormalities of Potential Clinical Concern
Description: Proportion (%) of participants with vital signs abnormalities (absolute and change from baseline) meeting categorical criteria over the 12-week double blind treatment period were counted. Vital signs data included blood pressure (BP) and pulse rate.
Time Frame: Week 4 to Week 16
Population: All participants who received any treatment during Week 4 (Visit 2) to Week 16 (Visit 5)
Measure: Number; unit: Percentage of Participants
Arm/Group | PF-05212377 30 mg | Placebo
Number analyzed (Participants) | 91 | 94
Percentage of Participants
  Absolute Supine Systolic BP<90 mmHg | 0 | 1.1
  Absolute Standing Systolic BP<90 mmHg | 0 | 1.1
  Absolute Supine Diastolic BP<50 mmHg | 0 | 2.1
  Absolute Standing Diastolic BP <50 mmHg | 0 | 0
  Absolute Supine Pulse Rate <40 bpm | 0 | 0
  Absolute Supine Pulse Rate >120 bpm | 0 | 0
  Absolute Standing Pulse Rate <40 bpm | 0 | 0
  Absolute Standing Pulse Rate >140 bpm | 0 | 0
  Increase in Supine Systolic BP>=30 mmHg | 0 | 5.3
  Increase in Standing Systolic BP>=30 mmHg | 2.2 | 3.2
  Increase in Supine Diastolic BP >=20 mmHg | 4.4 | 4.3
  Increase in Standing Diastolic BP >=20 mmHg | 3.3 | 5.3
  Decrease in Supine Systolic BP>=30 mmHg | 5.5 | 5.3
  Decrease in Standing Systolic BP>=30 mmHg | 5.5 | 5.3
  Decrease in Supine Diastolic BP >=20 mmHg | 8.8 | 5.3
  Decrease in Standing Diastolic BP >=20 mmHg | 4.4 | 6.4

24. Other Pre Specified Outcome: Participants in Each Category of C-CASA Mapped From the C-SSRS Responses
Description: Participants in each category of the Columbia Classification Algorithm of Suicide Assessment (C-CASA) mapped from the Columbia-Suicide Severity Rating Scale (C-SSRS) responses were reported.
  C-CASA Event Code: <1> Completed suicide; <2> Suicide attempt; <3> Preparatory acts towards imminent suicidal behavior; <4> Suicidal Ideation; <7> Self-injurious behavior, no suicidal intent.
  The suicidality assessments were performed at Screening, Week 0 (Visit 1), Week 4 (Visit 2), Week 6, (Visit 3), Week 10 (Visit 4), Week 16 (Visit 5), and Week 18 (Visit 6).
  Only participants falling any category of C-CASA events were listed below.
Time Frame: From Screening to Week 18/Early Termination
Population: All participants screened and assigned
Measure: Number; unit: Participants
Groups:
- Placebo Run-in: All participants assigned to the placebo run-in period
- Placebo: All participants received placebo during double blind period
Arm/Group | Placebo Run-in | PF-05212377 30 mg | Placebo
Number analyzed (Participants) | 195 | 91 | 94
Participants
  Week 4 (Visit 2): <4> | 1 | 2 | 1
  Week 6 (Visit 3): <4> | 0 | 0 | 1
  Week 10 (Visit 4): : <4> | 0 | 2 | 0
  Week 16/Early Termination (Visit 5): <4> | 0 | 1 | 0
  Week 4 (Visit 2): <7> | 0 | 0 | 1
  Week 6 (Visit 3): <7> | 0 | 1 | 0

ADVERSE EVENTS:
Time Frame: Baseline through Week 18 (Visit 16)
Groups:
- Placebo Run-In: Participants received placebo during the single blind placebo run-in period
Arm/Group | Placebo Run-In | PF-05212377 30 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 1/195 | 5/91 | 3/94
Other Adverse Events (participants affected / at risk) | 13/195 | 25/91 | 20/94
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Run-In (N=195) | PF-05212377 30 mg (N=91) | Placebo (N=94)
Bradycardia (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
Accidental death (General disorders) | 0 (0) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Foreign body (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Run-In (N=195) | PF-05212377 30 mg (N=91) | Placebo (N=94)
Diarrhoea (Gastrointestinal disorders) | 6 (6) | 8 (9) | 3 (3)
Urinary tract infection (Infections and infestations) | 0 (0) | 5 (5) | 4 (4)
Fatigue (General disorders) | 0 (0) | 2 (2) | 2 (2)
Bronchitis (Infections and infestations) | 0 (0) | 2 (2) | 1 (1)
Nasopharyngitis (Infections and infestations) | 4 (4) | 2 (2) | 2 (2)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 3 (3) | 3 (3)
Weight decreased (Investigations) | 1 (1) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1)
Hallucination (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.